CLINICAL TRIAL: NCT01512524
Title: Long Term Follow-up of Moderate and Severe Traumatic Bain Injury and Assessment of Involvement of Hormonal Deficiency in the Quality of Life
Brief Title: Hormonal Deficiency in the Quality of Life of Patients With Traumatic Brain Injury
Acronym: INSPIRE-TC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010.641
Record Dates: First submitted 2011-12-29; First posted 2012-01-19 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury (TBI)
Keywords: Traumatic Brain Injury; Quality of Life (QoL); hypopituitarism,GH
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients With Traumatic Brain Injury (Other): Study of the association between quality of life and MRI scans and endocrinology analysis (quantification of Growth Hormone) 18 months post-trauma.
  Interventions: Other: MRI scan and endocrinology analysis

INTERVENTIONS:
Other: MRI scan and endocrinology analysis — Endocrinology analysis including statique and dynamic exams, neuropsychologic evaluations and IRM scan.
  Other Names: MRI scan; endocrinology analysis

SUMMARY:
The primary objective is to assess the long-term impact of hormonal deficiency on Quality of Life (QoL) in a large group of moderate and severe Traumatic Brain Injury (TBI) patients.

DETAILED DESCRIPTION:
Severe Traumatic Brain Injury, when not leading to mortality, is a major cause of morbidity in early adulthood.

Recent studies have demonstrated a previously unappreciated association between Severe Traumatic Brain Injury and endocrine dysfunction.

The current trial aims at evaluating the quality of life 18 months post-trauma and associating this outcome to growth hormone levels.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be between the ages of 18-65
* Documented moderate to severe Traumatic Brain Injury (TBI) at less than 4 months post injury.
* Glasgow Coma Scale (GCS) equal to or greater than 12
* Patients volunteer to participate in the study, with a written informed consent signed
* BMI between 17 kg/m2 - 30kg/m2
* Affiliation to a national health insurance program

Exclusion Criteria:

* Glasgow Coma Scale (GCS) ≥13
* History of TBI ≥4 months
* Anterior hypopituitarism documented
* History of radiotherapy
* Liver dysfunction: total bilirubin <20µmol/l and/or factor V<60%)
* Renal dysfunction: creatinine clearance < 30 ml/mn (Cockcroft & Gault)
* Anyone who is currently taking or who has taken corticotherapy in the last 4 weeks before TBI
* Pregnancy
* Contraindications to MRI:
* Patients who have a heart pacemaker
* Patients who have a metallic foreign body (metal sliver) in their eye, or who have an aneurysm clip in their brain
* Patients with severe claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-11-23 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Evolution of the SF-36(Short-Form health survey)score up to 18 months post-trauma | assessed at 4 months (M4), 12 months (M12) and 18 months (M18) after brain injury.

SECONDARY OUTCOMES:
QOLIBRI (Quality of Life after Brain Injury) measure #1 | assessed at 4 months (M4), 12 months (M12)and 18 months (M18) after brain injury.
Questions on Life Satisfaction-Hypopituitarism (QLS-H) measure #2 | Time frame: assessed at 4 months (M4), 12 months (M12) and 18 months (M18) after brain injury.
Tests of Attentional, mnesic and executive performances #3 | assessed at 4 months (M4), 12 months (M12) and 18 months (M18) after brain injury.
  Tests of Attentional, mnesic and executive performances: - Alertness
  * Sustained Attention
  * Divided Attention
  * Go/NoGo
  * Working Memory
  * Incompatibility
  * Flexibility
  * Grober and Buschke test
  * Rey's complex figure (copy and memory)
Functional outcomes (#4):The Glasgow Outcome Scale (GOS)-Score | assessed at 4 months (M4), 12 months (M12) and 18 months (M18) after brain injury.
Functional outcome #5 :the Functional Independence Measure (FIM) | assessed at 4 months (M4), 12 months (M12) and 18 months (M18) after brain injury.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Courtois, MD, Principal Investigator — Hôpital Henry Gabrielle, Hospices Civils de Lyon
Locations (1):
- French University Hospital, Lyon, Auvergne-Rhône-Alpes, France